CLINICAL TRIAL: NCT06601179
Title: Phase 1-2 Dose-escalation Study, Evaluating the Safety and Efficacy of the "HIFU" High-intensity Focused Ultrasound Treatment of Benign Prostatic Hyperplasia After 3 Months, 6 Months, 12 Months, 18 Months and 36 Months.
Brief Title: Evaluating the Safety and Efficacy of the "HIFU" High-intensity Focused Ultrasound Treatment of Benign Prostatic Hyperplasia;
Acronym: BPH EFFICACY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU.F.23.02
Record Dates: First submitted 2024-07-08; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Phase 1 aims to determine the minimum effective dose for BPH treatment. It will include 10 patients receiving 50% of the standard shooting power. If, after a 3-month follow-up, there are no serious adverse events (SAEs) and good efficacy, Phase 2 will begin.
  If Phase 1 results indicate that 50% power is insufficient, power levels will be increased by 10% increments (60%, 70%, 80%, 90%) with similar follow-up until the minimum effective dose is determined.
  Phase 2 aims to validate the effocacy of the minimum effective dose. It will include 90 new patients treated with the same 50% power. They will be monitored regularly after 1 and 3 months, every 6 months up to 24 months, and finally at 36 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIFU (Experimental)
  Interventions: Device: HIFU

INTERVENTIONS:
Device: HIFU — high-intensity focused ultrasound treatment of benign prostatic hyperplasia

SUMMARY:
Prostate adenoma, also known as benign prostatic hypertrophy or hyperplasia (BPH), involves an increase in the size of the prostate, forming a benign tumor. It is the most common benign tumor in men, generally affecting those over 40 years old. The risk of BPH is more than 50% in men aged 50 to 60 and rises to 90% in men by age 80.

This hyperplasia leads to altered urinary flow and bladder outlet obstruction, referred to as "lower urinary tract symptoms" or LUTS, which become more frequent with age. These symptoms are categorized as obstructive or irritative. In the early stages, men with BPH may have difficulty starting urination and may feel as if their bladder is not completely empty. As a result, they need to urinate more often, especially at night, a condition known as nocturia. Additionally, the volume and velocity of the urinary flow may decrease significantly, as evidenced by flow measurements, and residual urine discharge may occur at the end of urination.

High-intensity focused ultrasound (HIFU) is a medical technique that uses high-intensity ultrasonic waves to treat various medical conditions, including malignant and benign tumors, without the need for invasive surgery or ionizing radiation. HIFU generates heat between 80° to 95°C at the focal point, causing necrosis of the targeted area with pinpoint accuracy. In urology, HIFU is used to treat prostate cancer in a minimally invasive manner, with focused ultrasounds delivered endorectally using a transducer that targets the treatment area with real-time monitoring.

Exclusively targeted HIFU treatment has been suggested for BPH, where localized necrosis of the side lobes reduces the volume of the prostatic transition zone, alleviating compression of the prostatic urethra and improving urinary symptoms.

This new study was initiated to evaluate the safety and efficacy of HIFU for BPH treatment.

ELIGIBILITY:
Inclusion Criteria:

Men aged ≥ 50 to ≤ 85

Patient diagnosed with benign prostatic hyperplasia evaluated by:

* Prostate volume ranging from 30 cc to 80 cc evaluated by MRI
* Qmax < 15ml/s
* IPSS ≥ 8
* IPSS-QoL ≥ 3
* IIEF-5 > 17

Patient for whom medical treatment failed (having been taken regularly for more than 12 weeks) OR patient with a contraindication to the initiation of medical treatment OR patient refusing medical treatment Patient whose prostate show no sign of cancerous lesion confirmed by MRI Patient capable of reading and understanding French or with a carer who speaks French and could help the patient understand the leaflet and the questionnaires Patient registered with a social security scheme Patient having given their free and informed consent to participate in the study

Exclusion Criteria:

Presence of a median lobe preventing the HIFU treatment to be delivered according to the investigator's judgment Prostate cancer confirmed or suspected History of surgical treatment of the prostate History of radiotherapy of the prostate History of bladder cancer History of urethral stricture Presence of a urinary tract fistula Urethral stricture or untreated bladder neck stenosis Untreated urinary lithiasis Neurological bladder or neurological bladder disease or any other neurological disease likely to affect the functioning of the bladder-sphincter system History of pelvic radiotherapy Patient with renal failure with GFR < 35ml/min Patient currently undergoing anticoagulant therapy (antivitamins K (AVK) and new oral anticoagulants (NOACs) for which the stop window cannot exceed 48H at the time of the HIFU procedure Contraindication to the surgical procedure, in particular anesthesia Contraindication to the pelvic MRI Patient with a rectal wall > 10mm

Contraindication to the HIFU treatment procedure:

* Active urogenital infection (the infection must be treated before HIFU treatment)
* Anal or rectal fibrosis, anal or rectal stenosis or any other abnormalities making it difficult to insert the Focal One® probe
* Urinary tract or rectal fistula
* Anatomic abnormalities of the rectum or rectal mucosa
* Presence of permanent radioactive implants in the rectal wall
* Presence of prostatic calcification the location of which interferes with the HIFU treatment
* Patient with an artificial sphincter, a penile prosthesis or intra-prostatic implant; for example, an endoprosthesis
* Presence of an implant (stent, catheter) within 1cm of the treatment area
* History of inflammatory bowel disease
* Presence of metal stents or implants in the urethra Patient refusing to participate in the study Person under guardianship considered legally incapable of giving their informed consentPatient unable or refusing to complete the questionnaires Persons placed under judicial protection Subject participating in another study including an exclusion period that is still running at the time of pre-inclusion

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | 3 months
  Phase 1
  Presence of significant cavitation that may be associated with adverse effects. Repeated urethral involvement that could damage the urethra. Absence of serious adverse effects (Clavien-Dindo ≥ III) directly attributable to the HIFU treatment procedure at 3 months of follow-up.
  Based on these elements, the scientific committee will analyze the cause-and-effect relationship between the indicators observed during treatment and the adverse effects.
Rate of patients with two of the following criteria ( Δ Qmax ≥ 50%, Δ IPSS ≥30%, Homogeneous necrosis observed on MRI) | 3 months
  Phase 1
  Efficacy :
  Efficacy will be considered satisfactory if at least two of the following three conditions are met:
  Significant improvement in the maximum flow defined by Δ Qmax ≥ 50% of the initial flow or by a removal of the urinary catheter or supra-pubic catheter in included patients with urinary retention.
  Improvement in obstructive and irritative symptoms 3 months after treatment, defined by a reduction in the IPSS score defined by Δ IPSS ≥30% Homogeneous necrosis observed on MRI
Rate of patients that meet the four evaluation criteria (Absence of AD Clavien-Dindo ≥ III + ΔQmax ≥ 50% + Δ IPSS ≥30% + IPSS-QoL score ≤2) | 6 months
  Phase 2
  Efficacy of the treatment
  To validate phase 2, 80% of patients are expected to meet the four evaluation criteria below after 6 months.
  Evaluation of urinary symptoms, continence, the erectile function, postoperative complications using a composite "tetrafecta" score defined by 4 criteria:
  1. Absence of serious adverse effects relating to the HIFU procedure, Clavien-Dindo ≥ III after 6 months.
  2. Significant improvement in the maximum flow defined by ΔQmax ≥ 50% of the initial flow after 6 months, or by a removal of the urinary catheter after 3 months in included patients with urinary retention.
  3. Improvement in obstructive and irritative symptoms 6 months after treatment, defined by a reduction in the IPSS score defined by Δ IPSS ≥30%
  4. Improvement in quality of life 6 months after treatment defined by an IPSS-QoL score ≤2

SECONDARY OUTCOMES:
Rate of adverse events | 36 months
  Treatment safety 1 month, 3 months, 6 months, 12 months, 18 months, 24 months and 36 months after treatment will be evaluated by:
  The rate of patients who experienced at least one adverse event with a Clavien-Dindo grade ≥ III The rate of patients with an SAE linked to the procedure The rate of patients with an SAE linked to the MD The rate of patients with unscheduled consultation and/or secondary re-hospitalization due to problems in connection with the procedure or the MD
Rate of patients with a significant decrease of prostate size | 36 months
  The impact of treatment on changes in prostate size will be evaluated by MRI and ultrasound 3 months, 6 months, 12 months after treatment.
The impact of the HIFU treatment on the urinary flow | 36 months
  The impact of the HIFU treatment on the urinary flow will be evaluated by measuring Q max 1 month, 3 months, 6 months, 12 months after treatment defined by:
  The rate of patient with ΔQmax ≥ 50% Rate of patients with removal of the urinary catheter after 3 months in included patients with urinary retention.
  The rate of patients with Qmax ≥ 15 ml/s
Rate of patients with a significant decrease of RPM | 36 months
  The impact of the HIFU treatment on bladder voiding will be evaluated by measuring RPM 1 month, 3 months, 6 months, 12 months after treatment, defined by:
  The rate of patients with RPM ≤ 150 ml The rate of patients with Δ RPM ≥50%
The rate of patients with a significant improvment of obstructive and irritative symptoms of the lower urinary tract | 36 months
  The effect of the treatment on the obstructive and irritative symptoms of the lower urinary tract will be evaluated using the IPSS score 1 month, 3 months, 6 months, 12 months, 24 months and 36 months after treatment, defined by:
  The rate of patients with Δ IPSS ≥30% The rate of patients with an IPSS score ≤ 7
The rate of patients with a significant improvment of LUTS-related quality of life | 36 months
  The evaluation of the impact of the HIFU treatment on LUTS-related quality of life 1 month, 3 months, 6 months, 12 months, 24 months and 36 months after treatment, defined by:
  The rate of patients with an IPSS-QoL score ≤ 2
The rate of patients with an improvment in the erectile function | 36 months
  The evaluation of the impact of treatment on the erectile function 1 month, 3 months, 6 months, 12 months and 36 months after treatment, defined by:
  The rate of patients with a Δ IIEF score ≤ 5
The evaluation of the impact of treatment on the ejaculatory function | 36 months
  The evaluation of the impact of treatment on the ejaculatory function 1 month, 3 months, 6 months, 12 months and 36 months after treatment, defined by:
  The rate of patients with a Δ MSHQ-EjD score < 25 The rate of patients with MSHQ-EJD <10 (no ejaculatory dysfunction or mild dysfunction) The rate of patients who say they suffer from retrograde ejaculation
The rate of patients with a recurrence over the follow-up period up to 36 months | 36 months
  The recurrence rate over the follow-up period up to 36 months will be evaluated by the number of patients with urinary retention who required catheterization or surgery for BPH.
The cost related to the use of HIFU | 36 months
  The estimation of costs related to the use of HIFU will be carried out by calculating the costs associated with consumables, the time of medical staff directly involved in the procedure, and the duration of hospitalization.
Efficiency | 36 months
  Efficiency will be estimated through the consideration of costs associated with HIFU treatment, follow-up costs, retreatments, and the duration of medical leave of absence.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Clinique Saint Vincent, Besançon
  - Clinique Tivoli-Ducos, Bordeaux
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU de Lille, Lille
  - HCL_Hôpital Edouard Herriot, Lyon
  - CH Matigues, Martigues
  - Hôpital Foch, Suresnes
  - Clinique Saint Michel, Toulon
  - Hôpitaux de Toulouse, Toulouse